CLINICAL TRIAL: NCT03916809
Title: Impact of Expiratory Muscle Strength Training (EMST) on Swallowing Function in Persons Undergoing Radiotherapy With or Without Chemotherapy (CRT) for Cancers of the Head and Neck (HNCA)
Brief Title: EMST in Patients Undergoing CRT for HNCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: Froedtert Hospital (Other); Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Barbara Pauloski, Associate Professor, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PRO29168
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Neoplasms; Deglutition Disorders
Keywords: oropharyngeal cancer; laryngeal cancer; swallow; chemoradiation; expiratory muscle strength training
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders; Oropharyngeal Neoplasms; Laryngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to an 8-week program of either Active Expiratory Muscle Strength Training (EMST) + Standard Care or Sham EMST + Standard Care in order to examine the impact of EMST on swallowing function.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will not know whether the device that they are given has a functioning valve spring or whether the valve spring has been removed.
  Researchers assessing the outcomes will not know the arm to which the subject was randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active EMST + Standard Care (Experimental): Patients randomized to the Active EMST + Standard Care arm (ACTIVE) will use the EMST150 device as packaged, i.e. following package instructions with a device that has its valve spring maintained.
  Interventions: Other: EMST
- Sham EMST + Standard Care (Sham Comparator): Those randomized to the Sham EMST + Standard Care arm (SHAM) will use an EMST150 device that has been modified by removing the internal spring, which allows the valve to open in response to airflow through the device regardless of the amount of pressure generated.
  Interventions: Other: EMST

INTERVENTIONS:
Other: EMST — Expiratory muscle strength training (EMST) is an exercise program designed to strengthen the muscles of expiration by increasing expiratory load during breathing exercises using either resistive or pressure threshold devices. The EMST150 is a commercially-available device considered non-significant risk (NSR). The EMST150 device will be used for this study.

SUMMARY:
This study is a randomized trial examining the impact of expiratory muscle strength training (EMST) on maintenance of safe and efficient oropharyngeal swallow function in persons with cancer of the head and neck (HNCA) undergoing treatment with radiation therapy or chemoradiotherapy (RT/CRT).

DETAILED DESCRIPTION:
Thirty (30) persons with newly-diagnosed HNCA who will be treated with RT/CRT will be randomized to an 8-week program of either Active Expiratory Muscle Strength Training (EMST) + Standard Care or Sham EMST + Standard Care in order to examine the impact of EMST on swallowing function. The training program will consist of 5 sets of 5 breaths, 5 days per week for 8 weeks, coincident with RT/CRT. Patients randomized to the Active EMST group will use the EMST150 (product name) expiratory muscle strength trainer according to package instructions. Those randomized to the Sham EMST group will use an EMST150 device that has been modified to eliminate resistance to airflow.

All subjects will be evaluated prior to initiation of cancer treatment (baseline assessment), 4 weeks into cancer treatment and again at the completion of cancer treatment (8 weeks after initiation of treatment). Assessment will include measurement of maximum expiratory pressure (MEP), a videofluoroscopic swallow study (VFSS) to objectively document swallow function, and administration of swallow-related quality of life (QOL) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of cancer in the oral cavity, oropharynx, hypopharynx, or larynx;
* Planned treatment with primary radiotherapy with or without chemotherapy;
* Age 18 or older and able to provide consent;
* Ability to use the EMST150 device (hold in mouth and maintain lip seal)

Exclusion Criteria:

* Primary surgery to the head and neck (neck dissection is permitted);
* Unknown primary tumor;
* Primary cancers of the nasopharynx, paranasal sinuses, salivary glands and skin.
* Progressive neurologic condition affecting muscle strength (e.g. amyotrophic lateral sclerosis (ALS), Parkinson's disease)
* Dysphagia not related to HNCA (e.g. unresolved swallowing difficulty post-stroke or post--traumatic brain injury (TBI))
* Prior history of head and neck radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-12 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Feeding-tube-free food intake (days) | 8 weeks
  the number of days from the beginning of the study until change in feeding status from 100% oral intake to combined oral intake and tube intake and/or 100% tube feeding will be calculated

SECONDARY OUTCOMES:
Penetration-Aspiration Scale rating (number) | 8 weeks
  From Videofluoroscopic Swallow Studies (VFSS), change in Penetration-Aspiration scale score will be determined from baseline to mid-treatment to post-treatment. Penetration-Aspiration Scale is an 8-point ordinal rating scale.
Timing of Aspiration (category) | 8 weeks
  From Videofluoroscopic Swallow Studies (VFSS), timing of aspiration will be determined from baseline to mid-treatment to post-treatment. Timing is identified as a category, either before, during, or after.
Presence of pharyngeal residue (dichotomous) | 8 weeks
  From Videofluoroscopic Swallow Studies (VFSS), the presence of residue in the pharynx (yes or no) will be determined from baseline to mid-treatment to post-treatment.
Extent of hyoid movement (mm) | 8 weeks
  From Videofluoroscopic Swallow Studies (VFSS), the change in extent of hyoid movement in mm will be determined from baseline to mid-treatment to post-treatment.
Upper esophageal sphincter (UES) opening width (mm) | 8 weeks
  From Videofluoroscopic Swallow Studies (VFSS), the change in width of UES opening width in mm will be determined from baseline to mid-treatment to post-treatment.

OTHER OUTCOMES:
Eating Assessment Tool (EAT-10) (number) | 8 weeks
  Change in score on the EAT-10 will be calculated from baseline to mid-treatment to post-treatment. EAT-10 is an ordinal rating scale with values that range from 0 to 40, with lower score reflecting better function.
M.D. Anderson Dysphagia Inventory (MDADI) (number) | 8 weeks
  Change in scores on the M.D. Anderson Dysphagia Inventory (MDADI) will be calculated from baseline to mid-treatment to post-treatment. MDADI consists of four ordinal rating scales with scores ranging from 0 to 100 with higher score reflecting better function.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pauloski, Principal Investigator — University of Wisconsin, Milwaukee
Locations (2):
- United States (2):
  - University of Wisconsin Milwaukee, Milwaukee, Wisconsin
  - Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No